CLINICAL TRIAL: NCT07373600
Title: Clinical and Radiographic Evaluation of Delayed Implant Placement Following Socket Preservation With Injectable Alloplastic Bone Graft. A Randomized Controlled Study.
Brief Title: Clinical and Radiographic Evaluation of Delayed Dental Implant Placement After Socket Preservation Using Injectable Bone Graft
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1004/2025
Record Dates: First submitted 2025-12-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Alveolar Ridge Preservation; Dental Implant Placement
Keywords: Dental Implant Placement; Alveolar Ridge Preservation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Extraction sites left to heal naturally without any bone grafting material before delayed implant placement. Dental implants will be placed after the natural healing period, and clinical and radiographic evaluations will be performed to assess ridge dimensions and implant outcomes
- Study Group (Experimental): Extraction sockets will be preserved using an injectable alloplastic bone graft material immediately after tooth extraction. After a healing period, delayed implant placement will be performed. Clinical and radiographic measurements will be used to evaluate ridge preservation and implant success.
  Interventions: Device: Injectable Alloplastic Bone Graft

INTERVENTIONS:
Device: Injectable Alloplastic Bone Graft — Following tooth extraction, socket preservation will be performed using an injectable alloplastic bone graft material composed of biocompatible synthetic components. The material will be placed into the extraction socket to maintain ridge dimensions and promote bone regeneration. After a healing period of several months, delayed implant placement will be performed, and clinical and radiographic evaluations will assess ridge preservation and implant success
  Arms: Study Group

SUMMARY:
This clinical study aims to evaluate the clinical and radiographic outcomes of delayed dental implant placement following socket preservation using an injectable alloplastic bone graft material.

The study will include patients who require tooth extraction and are candidates for implant placement.

After tooth extraction, the socket will be preserved using the bone graft material, and dental implants will be placed after a healing period.

Clinical and radiographic assessments will be performed to evaluate bone quality, bone height, and implant stability.

The goal of this study is to determine the effectiveness of injectable alloplastic bone grafts in maintaining the alveolar ridge and improving the success of delayed implant placement.

ELIGIBILITY:
* Patient aged between 40 and 60 years
* General good health.
* Volunteer subjects have to voluntarily sign an informed consent.
* Patient Indicated for single implant placement in lower posterior area.

Inclusion criteria for patients in group I

· Patient with a previously extracted lower posterior tooth and the socket was preserved with injectable bone graft .

Exclusion criteria:

* Patient with systemic disease affection bone metabolism .
* Patients with contraindication to surgical treatment.
* Patients with uncontrolled medical conditions.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Implant stability at the time of delayed implant placement | At the time of delayed implant placement (approximately 4 to 6 months after tooth extraction)
  Implant stability will be assessed at the time of delayed implant placement using resonance frequency analysis (RFA) to obtain implant stability quotient (ISQ) values. The ISQ readings will be used to evaluate the effect of socket preservation with injectable alloplastic bone graft on implant stability in comparison to sites without grafting.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT07373600/Prot_SAP_000.pdf